CLINICAL TRIAL: NCT02090738
Title: A Randomized, Open-label Study on Helicobacter Pylori Eradication With Standard Triple Regimen Plus Acetazolamide
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0941
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: H. Pylori Infection
MeSH Terms: interventions — Esomeprazole; BID protein, human; WW Domain-Containing Oxidoreductase; Amoxicillin; Clarithromycin; Acetazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm1 (Experimental): Treatment group
  Interventions: Drug: Acetazolamide group
- Arm2 (Active Comparator): Control group
  Interventions: Drug: Standard regimen group

INTERVENTIONS:
Drug: Acetazolamide group
  Other Names: Esomeprazole (Nexium®, AstraZeneca Korea, Co. Ltd., Seoul, Korea) 40 mg, bid, for 7 days; Amoxicillin (Kymoxin®, Yuhan Co. Ltd., Seoul, Korea) 1 g, bid, for 7 days; Clarithromycin (Klaricid®, Abbot Korea Co. Ltd., Seoul, Korea) 500 mg, bid, for 7 days; Acetazolamide (Diamox®, SK Chemicals Co. Ltd., Suwon, Korea) 250mg, bid, for 7 days
  Arms: Arm1
Drug: Standard regimen group
  Other Names: Esomeprazole (Nexium®, AstraZeneca Korea, Co. Ltd., Seoul, Korea) 40 mg, bid, for 7 days; Amoxicillin (Kymoxin®, Yuhan Co. Ltd., Seoul, Korea) 1 g, bid, for 7 days; Clarithromycin (Klaricid®, Abbot Korea Co. Ltd., Seoul, Korea) 500 mg, bid, for 7 days
  Arms: Arm2

SUMMARY:
Helicobacter pylori infection is associated with several gastric diseases, including gastritis, peptic and duodenal ulcers, gastric carcinoma and MALToma. In 1994, the WHO classified the organism as a type 1 carcinogen. In order to eradicate H. pylori, at least two antibiotics and a proton pump inhibitor are used as a standard therapy regimen. Emerging antibiotic resistance to metronidazole or clarithromycin, however, has made successful treatment of infection progressively more difficult, with the success rate of standard triple therapy now at 70%, well below the 80% required for treatment of infectious diseases. Therefore, new treatment regimen is required for successful H. pylori eradication.

On the other hands, many in vitro studies revealed that bacterial carbonic anhydrase in H. pylori has an important role for surviving of H. pylori in the stomach. It was demonstrated that mutation of carbonic anhydrase affected survival of H. pylori. The investigators therefore expected that administration of carbonic anhydrase inhibitor (acetazolamide) with standard H. pylori eradication regimen would increase the eradication rate. Here, the investigators aim to evaluate the efficacy of standard triple regimen plus acetazolamide for H. pylori eradication.

ELIGIBILITY:
Inclusion Criteria:

1. Age, between 19 and 70
2. H. pylori infected patients

Exclusion Criteria:

1. Previous history of H. pylori eradication
2. Previous history of gastrectomy
3. Administration of PPI, H2 blocker, antibiotics, or bismuth within 1 month prior to enrollment
4. Allergy to sulfonamide
5. Electrolyte imbalance
6. Adrenal insufficiency
7. Pregnancy or breast milk feeding
8. Active infection
9. Severe hepatic dysfunction
10. Severe renal dysfunction
11. Severe bone marrow dysfunction
12. Significant neurologic or psychologic disease

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rate | 1 month from the eradication therapy
  H. pylori eradication rate will be assessed by urea breath test after eradication therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- severnace Hospital, Seoul, Seodaemun-gu, South Korea